CLINICAL TRIAL: NCT03006952
Title: Comparative Effects of add-on Pentoxifylline to Losartan Versus Increasing Dose of Losartan on Serum NT-PRO BNP and Proteinuria in Type 2 Diabetics With Nephropathy
Brief Title: Add-on Pentoxifylline to Losartan Versus Increasing Dose of Losartan on NT-PRO BNP in Type 2 Diabetics With Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 931133003
Record Dates: First submitted 2016-12-24; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Pentoxifylline; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pentoxifylline & losartan (Active Comparator): pentoxifylline arm took 400 mg pentoxifylline twice daily plus 50mg losartan daily for 12 weeks.
  Interventions: Drug: Pentoxifylline; Drug: Losartan
- Losartan (Active Comparator): losartan arm took 100mg losartan daily for 12 weeks.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Pentoxifylline — pentoxifylline arm took 400 mg pentoxifylline twice daily plus 50mg losartan daily for 12 weeks.
  Other Names: oxpentifylline
  Arms: pentoxifylline & losartan
Drug: Losartan — losartan arm took 100mg losartan daily for 12 weeks.
  Other Names: Cozaar

SUMMARY:
This study was designed to assess the efficacy of adding pentoxifylline to losartan in comparison with increasing dose of losartan in type 2 diabetes patients with nephropathy. also the effect of pentoxifylline on N terminal brain natriuretic peptide (NT-pro BNP) and C-reactive protein

DETAILED DESCRIPTION:
Addition of pentoxifylline to losartan provides antiproteinuric effects in type 2 diabetes patients with nephropathy that might relate to its effect on N terminal brain natriuretic peptide (NT-pro BNP) and C-reactive protein.

Pentoxifylline is a phosphodiestrase inhibitor with anti-inflammatory effects that was used in type 2 diabetes patients with nephropathy for treatment of diabetes complications.

NT-Pro BNP, which is released from the heart due to wall stress and pressures, is known as a diagnostic and prognostic marker for heart failure and cardiovascular mortality in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age>30 and age<70, urinary albumin excretion (UAE) ≥150 mg/24 h

Exclusion Criteria:

* any infectious or malignant diseases, non-diabetic kidney disease, retinal hemorrhage, acute myocardial infarction, uncontrolled hypertension, pregnancy, unable to follow up, hyperthyroidism, baseline serum potassium concentrations ≥5.5 meq/L, glomerular filtration rate (GFR)<30mL/min/1.73 m and intolerance of pentoxifylline

Ages: 38 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
N terminal brain natriuretic peptide (NT-pro BNP) | 3 months
  N terminal brain natriuretic peptide assessed using ELISA method (zelbio, Germany) with inter- and intra-assay coefficient of variation (CV) <12% and <10%. Measured at baseline, 3rd month

SECONDARY OUTCOMES:
Highly sensitive C-reactive protein (hsCRP) | 3 months
  Highly sensitive C-reactive protein assessed by commercial kits (DRG kit, Germany) using the ELISA (enzyme-linked immunosorbent assay) method with inter- and intra-assay coefficient of variation (CV) of <20%. Measured at baseline, 3rd month
Urinary albumin excretion | 3 months
  Urinary albumin excretion assessed by overnight (12 hour) collection of urine. Measured at baseline, 3rd month
Blood pressure | 3 months
  Systolic and diastolic blood pressure assessed by mercury sphygnomanometry. Patients were placed in a sitting position and after ten minutes rest, two readings from right-side hand with five minutes interval were obtained. Measured at baseline, 3rd month
estimated glomerular filtration rate | 3 months
  estimated glomerular filtration rate calculated using the formula developed by Chronic Kidney Disease Epidemiology Collaboration. Measured at baseline, 3rd month
serum creatinine concentrations | 3 months
  serum creatinine concentrations assessed by Jaffe method. Measured at baseline, 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, MD, Study Chair — Endocrinology and Metabolism Research Center (EMRC), Vali-Asr Hospital, Tehran University of Medical Sciences, Tehran, Iran
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes